CLINICAL TRIAL: NCT07363655
Title: Effects of a Rehabilitation Programme Focused on Energy Management in People With Myalgic Encephalomyelitis / Chronic Fatigue Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Saúde Norte da Cruz Vermelha Portuguesa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024.063
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Myalgic Encephalomyelitis (ME); Chronic Fatigue Syndrome (CFS)
Keywords: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS);; energy management;; pacing; fatigue; physical function; quality of 19 life.)
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — An educational program focused on energy management and developed by the United Kingdom's NICE. The overall aim of the intervention was the empowerment of patients with self-management strategies that could help them to maximize their autonomy, independence and daily activities without exceeding their perceived energy reservoir.

SUMMARY:
The study focuses on rehabilitation nursing care for adults diagnosed with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome in a home setting. The objective is to evaluate the effects of an individualised rehabilitation programme, which aims to empower participants to manage their energy effectively, observing the impacts on functionality and fatigue.

DETAILED DESCRIPTION:
During the study, we collected sociodemographic data, information about the clinical evolution, patient perception of the disease. Instruments were applied to assess quality of life, functionality, and fatigue levels. This will allow to understand how to improve rehabilitation nursing care.

ELIGIBILITY:
Inclusion Criteria:

* Portuguese-speaking individuals with age of 18 years or older;
* Individuals with official residence in Portugal;
* An official diagnosis of ME/CFS based on the NICE guidelines;
* A Chalder's Fatigue Questionnaire (CFQ) score higher than 18 points.

Exclusion Criteria:

* Individuals without official residence in Portugal;
* Patients without a diagnosis of ME/CFS;
* Patients with a diagnosis of ME/CFS whose case definitions used was not known;
* Patients without a diagnosis of ME/CFS who had previously participated in any kind of rehabilitation programme, including pacing therapy, cognitive behavioural therapy or graded-exercise therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-03-09 (Actual)

PRIMARY OUTCOMES:
Functional Assessment | Assessment at two time points: M0 - before the start of the intervention; M1 - 12 weeks after the end of the intervention.
  Short Form Health Survey: SF 36 v2 (physical dimension)
Quality of Life Measure | Assessment at two time points: M0 - before the start of the intervention; M1 - 12 weeks after the end of the intervention.
  Quality-of-life measure: EuroQoL 5D-5L
Fatigue Assessment | Assessment at two time points: M0 - before the start of the intervention; M1 - 12 weeks after the end of the intervention.
  Application of the Chalder Fatigue Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde Norte da Cruz Vermelha Portuguesa, Portugal., Oliveira de Azeméis, Aveiro District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided